CLINICAL TRIAL: NCT00886418
Title: Effect of Continuous Myorelaxation on the Need for Hypnotic Agent During Surgical Procedures Which do Not Require it (Multicenter, Randomized and Prospective Study)
Brief Title: Influence of Muscle Relaxation on a Closed-loop Anesthesia System
Acronym: Drone-Curare
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/28
Record Dates: First submitted 2009-04-19; First posted 2009-04-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Total intravenous anesthesia (propofol and remifentanil) is provided using the close-loop system. A muscle relaxant is used to facilitate tracheal intubation; its administration is continued throughout anesthesia.
  Interventions: Drug: muscle relaxant
- 2 (Experimental): Total intravenous anesthesia (propofol and remifentanil) is provided using the close-loop system. No muscle relaxant is used and a placebo is infused throughout anesthesia.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: muscle relaxant — muscle relaxant administration throughout anesthesia
  Arms: 1
Drug: normal saline — no muscle relaxant throughout anesthesia (normal saline infused as a placebo)
  Arms: 2

SUMMARY:
Total intra-venous anesthesia can be provided using a closed-loop system guided by the bispectral index. The purpose of this study is to determine if myorelaxation modifies its functioning.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for a surgical procedure which not require a myorelaxation

Exclusion Criteria:

* age less than 18 years,
* ASA III and above,
* pregnant woman
* combined general and regional anesthesia,
* history of prolonged myorelaxation due to a decrease in cholinesterase,
* patient with a known lack in cholinesterase,
* history of cerebral or psychiatric central,
* allergy to latex, propofol, remifentanil, morphine, muscle relaxant or any of the excipients,
* known hypersensitivity to remifentanil or to an other derivative of fentanyl,
* presence of a pacemaker,
* psychotropic or agonist-antagonist morphine treatment,
* planned post-operative sedation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
propofol dose | one hour anesthesia

SECONDARY OUTCOMES:
remifentanil dose | one hour anesthesia
number of automatic modifications of the propofol and remifentanil concentrations | one hour anesthesia
number of patients' movements | one hour anesthesia
number of hemodynamic abnormalities requiring treatment | one hour anesthesia
time to wake up | end of anesthesia
intraoperative awareness | postoperative day 1 or 2
performance of the closed-loop system | one hour anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (3):
- France (3):
  - CHU Besançon, Besançon
  - Institut Paoli-Calmette, Marseille
  - Hôpital Foch, Suresnes